CLINICAL TRIAL: NCT03484195
Title: Neoadjuvant FOLFOXIRI (Irinotecan, Oxaliplatin and Fluorouracil) Chemotherapy in Patients With Locally Advanced Colon Cancer：an Open-label, Single-arm, Multicenter Phase II Study
Brief Title: Neoadjuvant FOLFOXIRI Chemotherapy in Patients With Locally Advanced Colon Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Director, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGIOG-2017-01
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Colonic Neoplasms; Drug Therapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — FOLFOXIRI protocol; Irinotecan; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOXIRI (Experimental): Patients received 4 cycles of neoadjuvant FOLFOXIRI chemotherapy before surgical resection.
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI — Irinotecan 150 mg/m^2 IV over 1h, day 1 + Oxaliplatin 85 mg/m^2 IV over 2h, day 1 + L-Leucovorin 200 mg/m^2 IV over 2h, day 1 + 5-Fluorouracil 2800 mg/m^2 IV 48h continuous infusion, starting on day 1 administered every two weeks for 4 cycles (2 months)
  Other Names: Irinotecan; Oxaliplatin; 5-Fluorouracil

SUMMARY:
To evaluate the efficacy and safety of neoadjuvant FOLFOXIRI chemotherapy (irinotecan, oxaliplatin and fluorouracil) in the patients with locally advanced colon cancer.

DETAILED DESCRIPTION:
For the patients with locally advanced colon cancer, adjuvant FOLFOX and XELOX chemotherapy have become standard treatment. However, 30% - 40% patients suffered from local recurrence or distant metastasis after this standard treatment. Neoadjuvant chemotherapy could shrink tumors, eliminate micrometastasis, reduce surgical trauma and accelerate recovery. Hence, we evaluate the efficacy and safety of FOLFOXIRI as neoadjuvant chemotherapy in treating patients with locally advanced colon cancer.

In this prospective study, 30 patients with locally advanced colon cancer will be treated with 4 cycles of neoadjuvant FOLFOXIRI chemotherapy followed by surgical resection. PET-CT scanning will be performed before and after the neoadjuvant FOLFOXIRI chemotherapy to assess SUVmax changes. The ctDNA in peripheral blood before and after each cycle of neoadjuvant FOLFOXIRI chemotherapy will be detected. In the course of treatment, safety evaluation will be carried out according to adverse reaction classification (CTCAE) 4. 0.

ELIGIBILITY:
Inclusion Criteria

* Age: 18-75years old
* Primary and pathological diagnosis of colon adenocarcinoma
* Radiographic evaluation of initial resectable colon cancer
* T4b colon cancer
* ECOG status: 0～1
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

Neutrophil count≥1.5×10^9/L Platelet count≥90×10^9/L Hemoglobin≥90g/L Total bilirubin (TBI) ≤ 1.5 * ULN Alanine aminotransferase (ALT)≤2.5 * ULN Aspartate aminotransferase (AST)≤2.5 * ULN Alkaline phosphatase (ALP)≤2.5 * ULN

* Signed informed consent; able to comply with study and/or follow- up procedures

Exclusion Criteria:

* Previous treatment with oxaliplatin, irinotecan or fluorouracil
* Hypersensitivity to fluorouracil, oxaliplatin or irinotecan.
* With distant metastasis
* Cardiovascular disease that would preclude study treatment or follow-up; New York Heart Association class III or IV heart disease; active ischemic heart disease; myocardial infarction within the past 6 months; symptomatic arrhythmia uncontrolled hypertension. Unexplained syncope occurred within 3 months
* Digestive system diseases that would preclude study treatment or follow-up within the past 6 months
* Gastric ulcers or duodenal ulcers for the treatment of resistance;
* 3 or 4 grade gastrointestinal bleeding / bleeding;
* Gastrointestinal perforation / fistula;
* abdominal abscess;
* Infectious or inflammatory bowel disease
* HIV infection and/or active hepatitis B virus infection
* Pregnant or lactating women. Fertile patients must use effective contraception
* Any serious acute or chronic disease that can not be involved in the study or to influence the interpretation of the results of the study
* Other intervention clinical trials were combined at the same time.
* Nerve or mental abnormality affecting cognitive ability
* Other malignancy except effectively treated squamous cell or basal cell skin cancer,
* Other situations that the researchers think should be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
The ratio of tumor downstaging to stage 0 and stage I | 2 years
  Tumor downstaging from stage II or III to pathologic complete response (stage 0) and stage I

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | 2 years
  The level of tumor regression under pathological examination
Disease free survival | 3 years
  Estimated from the date of surgery to the date of recurrence
Overall survival time | 3 years
  Estimated from the date of enrollment to death from any cause
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 years
  The grade of toxicity will be assessed using the NCI-CTCAE version 4.0
ctDNA change | 3 years
  The relationship between ctDNA and survival will be evaluated
SUVmax changes | At the begin of Cycle 1 and the end of Cycle 4 (each cycle is 14 days)
  Tumor metabolic response through FDG-PET examination before and after 4 cycles of neoadjuvant FOLFOXIRI chemotherapy
Quality of life (QLQ C30) | Every 2 weeks after the first treatment until 3 years
  Scores according to EORTC QLQ-C30 scoring manual

CONTACTS AND LOCATIONS:
Overall Officials: Jingdong Zhang, Study Chair — Cancer Hospital of China Medical University, Department of Medical Oncology, Liaoning Cancer Hospital & Institute
Locations (1):
- Liaoning Cancer Hospital, Shenyang, Liaoning, China